CLINICAL TRIAL: NCT01427400
Title: The Use of Botulinum Toxin-A in Two-stage Tissue Expander/Implant Breast Reconstruction: A Prospective, Randomized, Double-Blind Placebo Controlled Trial
Brief Title: The Use of Botulinum Toxin A in Two-Stage Tissue Expander/ Implant Breast Reconstruction
Acronym: Botox
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government); Providence Health & Services (Other); Fraser Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H10-03166
Record Dates: First submitted 2011-08-18; First posted 2011-09-01 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases
Keywords: Breast expander; Breast reconstruction; Implants; Botox
MeSH Terms: conditions — Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expander Placement, Botulinum Toxin-A (Experimental): During surgery, administered only once, 5 cc in 5 different locations on chest muscle.
  Interventions: Drug: Botulinum Toxin-A
- Tissue expander Placement WITH Saline (Placebo Comparator): During surgery, administered only once, 5 cc in 5 different locations on chest muscle.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Botulinum Toxin-A — 100 Units diluted in 25cc saline
  Other Names: Botulinum Toxin Type A
  Arms: Expander Placement, Botulinum Toxin-A
Drug: Saline — Dispensed in a 25cc syringe
  Other Names: 0.9% Sodium Chloride
  Arms: Tissue expander Placement WITH Saline

SUMMARY:
Breast reconstruction is a common procedure with over 86,000 breast reconstruction procedures performed in the United States in 2009. This is a 1.5-fold increase since 2007. Of these breast reconstructions, 65% use a tissue expander/implant technique. Although satisfactory results can be achieved with a single-stage technique, a two-stage approach is considered more reliable, allowing for precise positioning of the inframammary fold and an opportune time to perform a capsulotomy to increase the breast skin flap by releasing the soft tissue.

The placement of the tissue expander and implant under the chest muscles is thought to minimize the incidence of capsular contracture, expander exposure, and in addition, produce acceptable aesthetic results. However, discomfort is often associated with this submuscular placement of a tissue expander or implant, specifically during the expansion phase. Patients undergoing immediate reconstruction using submuscular implants have been shown to have higher analgesic requirements and to have higher pain scores post-operatively, compared to non-reconstructed patients. An uncomfortable reconstruction can lead to under-filling of the expander, a longer expansion process, abandonment of reconstruction, and a compromised quality of life. The use of Botulinum Toxin A (Botox) injections into the chest muscles at the time of surgery may help ease the discomfort that is often associated with this procedure.

The investigators propose a prospective double-blind randomized placebo-controlled trial of patients undergoing tissue expander/implant reconstruction. The information gathered from this analysis will provide a greater understanding of the effects of Botox in the setting of two-stage tissue expander/implant breast reconstruction, with the goal to improve patient satisfaction and quality of life.

DETAILED DESCRIPTION:
Currently, there is level C evidence for the efficacy of Botox in the treatment of postoperative pain and muscle spasms in breast reconstruction patients. Additional high-level evidence is necessary to justify the use of Botox in breast cancer patients, which potentially will improve the reconstructive process for these patients and improve quality of life. Additionally, there have been no studies to date that have evaluated patient satisfaction and QOL in this setting. The investigators will evaluate patient satisfaction and QOL using the Breast-Q© during different time periods after two-stage tissue expander/implant reconstruction. Previous studies have demonstrated a reduction in pain when Botox was used during tissue expander/implant breast reconstruction, however, these studies were not blinded which may introduce bias. Additionally, a timely reconstruction is important to the patient, and a decrease in pain may result in a shorter fill interval and an increased total amount of volume in the tissue expander. The investigators will therefore document both the amount of expansion that a patient can tolerate at each follow-up visit and the total volume expanded, and compare the data between the Botox group to the group assigned to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo immediate, post-mastectomy, unilateral or bilateral, tissue expander/implant reconstruction
* Patients older than 21, with no upper age limit
* English-speaking, or has an appropriate translator

Exclusion Criteria:

* Patient declines inclusion in the study
* Patients who undergo a single-stage implant reconstruction or combined autogenous tissue expander/implant reconstruction
* Previous history of radiation
* Previous breast surgery with implants
* Previous history of axillary lymph node dissection
* Patients who are pregnant
* Patients with hepatorenal failure
* Patients with known hypersensitivity to Botulinum Toxin-A
* Patients with significant mastectomy flap ischemia at time of tissue expander placement

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Quality of life and patient satisfaction using the Breast-Q | Before 1st surgery, 2 weeks, ~6-8weeks, Before 2nd Surgery, 6 months, and 12 months post-op
  The Breast-Q© is a patient reported outcome measure (PROM) for breast surgery that was rigorously developed to accurately measure patient reported satisfaction and quality of life (QOL). (http://www.mskcc.org/mskcc/shared/Breast-Q/index.html). The BREAST-Q was developed and validated with adherence to international guidelines. This PROM is composed of six scales that address: 1) psychosocial well-being, 2) physical well-being, 3) sexual well-being, 4) satisfaction with breasts, 5) satisfaction with outcome, and 6) satisfaction with care.

SECONDARY OUTCOMES:
Patient-reported pain,using the BPI (Brief Pain Inventory) and Pain Diary during the expansion phase (initial to final expansion) and in the long-term period (6 and 12 months). | BPI (before 1st surgery, day of surgery, 2 weeks, ~ 6 - 8 weeks, before 2nd surgery, 6 months and 12 months). After 1st surgery, pain diary is to be filled out every evening at the same time.
  The BPI is a common patient-reported instrument used to assess clinical pain. The BPI assesses the severity of pain and the impact of pain on daily functions in patients with pain from chronic diseases or conditions or acute conditions (i.e. postoperative pain).
  The question asked on the daily pain diary will be derived from the BPI: "Every evening at the same time, please rate the worst pain you've experienced in the last 24 hours when 0 represents no pain and 10 represents the most severe pain imaginable".
Aesthetic outcome | 6 months and 12 months (after 2nd surgery)
  Aesthetic results can be evaluated using different methods: patient-reported aesthetic satisfaction (Breast-Q) and aesthetic outcome from the perspective of the health professional. Standardized photographs using a three-category, five-item Breast Aesthetic Score. This scoring scheme separates the various components of the aesthetic results of the breast into different subscale thus allowing the rating to be more explicit. This score has not been validated, but has demonstrated good inter- and intra-rater reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Adelyn Ho, MD, MPH, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Plastic, Reconstructive and Cosmetic Surgery, Surrey, British Columbia
  - Canada, British Columbia, Vancouver, British Columbia

REFERENCES:
- See also: UBC Division of Plastic Surgery — http://www.surgery.ubc.ca/plasticsurg.html
- See also: Canadian Breast Cancer Foundation — http://www.cbcf.org